CLINICAL TRIAL: NCT04134754
Title: The Role of Central CO2 Chemosensitivity in Postictal Respiratory Depression and SUDEP
Brief Title: Carbon Dioxide (CO2) Chemosensitivity and SUDEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brian Gehlbach, MD, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201908728; 1R01NS113764-01 (NIH)
Record Dates: First submitted 2019-10-08; First posted 2019-10-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy; SUDEP
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy

STUDY DESIGN:
Intervention Model Description: Basic Experimental Studies in Humans (BESH)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Respiratory physiology testing (Other): Subjects will wear a nosepiece and breathe through a Y-valve that allows switching from room air to two 5-liter rebreathing bags pre-filled with 50% O2, 6% CO2, and balance N2. Ventilation and respiratory gases will be measured using a pneumotachograph and rapid gas analyzers (Ultima PFX pulmonary function/stress testing system, Medical Graphics Corp). In subjects who experience clinical seizure-like activity, we will repeat the HCVR. This repeat test will occur 2 or more hours after a generalized convulsive seizure (GCS). We will repeat the HCVR at least 30 minutes after a non-GCS. Finally, we may repeat the HCVR at least 18 hours after the last seizure (GCS or non-GCS). It is anticipated that some subjects may exhibit frequent seizures that necessitate the adjustment of this schedule. Subjects may also be asked to sniff, hold their breath, and breathe through tubes of different sizes.
  Interventions: Other: 6% Carbon dioxide/50% oxygen/balance nitrogen mixture

INTERVENTIONS:
Other: 6% Carbon dioxide/50% oxygen/balance nitrogen mixture — In the hypercapnic ventilatory response (HCVR) test, the subject will rebreathe a gas mixture that has 6% carbon dioxide and 50% oxygen. This test has been performed for decades for research and clinical purposes. The effects of carbon dioxide inhalation are short lived and do not cause long term consequences. the hypercapnic ventilatory response (HCVR), we will have you

SUMMARY:
The purpose of this research study is to better understand what causes Sudden Unexpected Death in Epilepsy (SUDEP). This study will enroll subjects from the University of Iowa Hospitals and Clinics (UIHC) Epilepsy Monitoring Unit (EMU) and Epilepsy Clinics. The investigators will analyze the effects of seizures on breathing, on the cardiovascular system, and on arousal. The investigators are studying these effects because some cases of SUDEP might be due, in part, to an inability to wake up or sense elevated carbon dioxide (CO2) levels when breathing is impaired. Subjects will be followed for ten years after enrollment to monitor their health.

DETAILED DESCRIPTION:
In this study, the investigators will only enroll adults with confirmed or suspected epilepsy; there is no control group. Patients admitted to the UIHC Epilepsy Monitoring Unit (EMU) for continuous VideoEEG will undergo video recordings of their face and body, electroencephalography (EEG), and electrocardiogram (ECG) as part of their normal clinical care. Research subjects will undergo noninvasive cardiorespiratory monitoring during their EMU stay for the purpose of correlating heart rate and breathing patterns with EEG patterns related to their seizures.

Eligible subjects will undergo several respiratory tests. This may include sniffing and breath holding and breathing through tubes of different sizes. One test, called the hypercapnic ventilatory response (HCVR), will have you rebreathe a gas mixture of 6% carbon dioxide and 50% oxygen to look at how more you breath in response to the increase in carbon dioxide levels. The investigators will then measure how much more subjects breathe in response to the increase in carbon dioxide levels, and also how breathing feels at the end of the test. The investigators will analyze the relationship between the HCVR and cardiorespiratory changes from seizures. The investigators will also analyze the effect of seizures on the HCVR. The HCVR test will be done by our respiratory therapist during subjects' stay in the EMU.

Some subjects will be asked to participate in repeat testing of the HCVR 3 more times as an outpatient over the next 2 years. Additional subjects will also be enrolled from the clinic and will also undergo HCVR testing 4 times over the 2 years. All subjects will agree to undergo an interview in person or by phone, email, or questionnaire annually for ten years. They will also provide consent for follow-up with a personal contact in the event of subject death, for the purpose of ascertaining whether the death was due to SUDEP.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is between 18 and 99 years of age.
2. Confirmed or suspected epilepsy.
3. Admission to the EMU for spell characterization (EMU group) or undergoing care in the University of Iowa Health Care Epilepsy Clinic.

Exclusion Criteria:

1. History of uncontrolled cardiac, pulmonary, or hepatic disease.
2. Progressive or uncontrolled neurologic disease unrelated to epilepsy.
3. Current opioid use.
4. Women of child-bearing potential who are pregnant or capable of becoming pregnant (e.g. sexual activity within the past 21 days without a highly effective form of birth control or positive urine pregnancy test).
5. Other comorbid condition that may influence the safety or feasibility of HCVR testing.
6. Limited decision-making capacity and absence of a qualified representative.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Determine the correlation between baseline central CO2 chemosensitivity and the increase in transcutaneous CO2 levels after a seizure. | Immediately before and after a seizure, variable for each subject but approximately 10 minutes
  The change in HCVR slope (change in minute ventilation [liters/min] vs change in end tidal CO2 [mm Hg]) will be correlated with the increase in transcutaneous CO2 level (mm Hg) provoked by a seizure.
Determine the correlation between baseline central CO2 chemosensitivity and the duration of transcutaneous CO2 elevation above baseline after a seizure. | Duration of hospital admission, approximately 5 days
  The change in HCVR slope (change in minute ventilation [liters/min] vs change in end tidal CO2 [mm Hg]) will be correlated with the duration (minutes) of end tidal CO2 elevation above pre-seizure baseline
Effect of seizures on HCVR slope (liters/min/mm Hg) | Up to 18 hours after a seizure.
  The percent change in HCVR slope (liters/min/mm Hg) from baseline that is induced by a seizure will be measured. The HCVR will be administered at 30 minutes, 2 hours, and 18 hours after nonconvulsive seizures. The HCVR will be administered at 2 hours and 18 hours after convulsive seizures.
Determine the stability of the HCVR slope over time in patients with epilepsy. of the HCVR over time in patients with epilepsy | 2 years
  The stability of the HCVR slope (liters/min/mm Hg) measured 8 months for 2 years will be assessed using a generalized linear mixed model.

SECONDARY OUTCOMES:
Change in respiratory rate provoked by seizures | Immediately before and after a seizure, variable for each subject but approximately 10 minutes
  Frequency of breaths (breaths/minute) will be measured using respiratory effort belts around the chest and abdomen

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gehlbach, MD, Principal Investigator — University of Iowa; George Richerson, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared upon with qualified investigators upon completion of the study, under the guidelines of the NIH Data Sharing Policy and Implementation Guidance and under the control of the Principal Investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data elements will be potentially eligible for sharing 1 year after the study has been completed and the results have been disseminated via a summary report.
Access Criteria: Direct communication with the Principle Investigators.